## **Cover Page for the Data Analysis Plan**

| Official Title: | Mobile health (mHealth) application called CBCT Sessions to Treat and Reduce Elevated Stress among Students (C-STRESS) |
|---|---|
| NCT Number: | NCT05776901 |
| Document Type: | Data Analysis Plan |
| Document Date: | 08/09/2023 |

## **C-STRESS Statistical Analysis Plan**

The primary outcome will be C-STRESS's usability as reflected in usability scores and measured by the System Usability Scale (SUS). Descriptive statistics (i.e., mean and standard deviation) of the usability scores of the C-STRESS platform at the baseline, week 3, and week 6 will be computed. Two-sided, paired-sample t-tests will be used to evaluate the change in mean SUS scores from baseline at week 3 and week 6.